CLINICAL TRIAL: NCT05711524
Title: Pilot Clinical Trial of Transfusion of Pathogen Reduced Cryoprecipitated Fibrinogen (INTERCEPT Fibrinogen Complex) in Patients With Bleeding to Expedite Product Availability and Improve Outcomes in Perioperative Bleeding
Brief Title: Transfusion of Pathogen Reduced Cryoprecipitated Fibrinogen to Expedite Product Availability in Perioperative Bleeding
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Cerus Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-04024649
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Hypofibrinogenemia; Bleeding
Keywords: Cryoprecipitate; Pathogen Reduced Cryoprecipitate
MeSH Terms: conditions — Afibrinogenemia; Hemorrhage

STUDY DESIGN:
Intervention Model Description: The intervention and randomization are not made at the level of the individual patient, but rather on clusters of patients by month. The clusters will include all patients at NYP/WC for whom pooled cryo is ordered during a single month.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients given Traditional Cryo (Active Comparator): These are the liver transplant and cardiothoracic (LT and CT) patients that will be given traditional cryo based on the randomization protocol. The blood bank will alternate use of PR cryo and regular cryo each month for all patients with a cryo order. All patients will receive either traditional cryo or PR cryo in a given month.
  Interventions: Biological: Traditional Cryoprecipitate
- Patients given PR Cryo (Experimental): These are the liver transplant and cardiothoracic (LT and CT) patients that will be given PR cryo based on the randomization protocol. The blood bank will alternate use of PR cryo and regular cryo each month for all patients with a cryo order. All patients will receive either traditional cryo or PR cryo in a given month.
  Interventions: Biological: Pathogen-Reduced Cryoprecipitate

INTERVENTIONS:
Biological: Traditional Cryoprecipitate — This is the cryoprecipitate already currently being given to patients with a cryo order.
  Arms: Patients given Traditional Cryo
Biological: Pathogen-Reduced Cryoprecipitate — This is the pathogen-reduced cryoprecipitate that is intended to be compared to the standard cryoprecipitate.
  Arms: Patients given PR Cryo

SUMMARY:
The goal of this quality improvement study is to compare pathogen-reduced cryoprecipitate with traditional cryoprecipitate in liver transplant and cardiovascular patients. The investigators hypothesize that by having immediate access to a readily available thawed blood product that replaces fibrinogen (the main substrate of a blood clot), early bleeding can be treated before it escalates into uncontrolled hemorrhage, and therefore additional blood products, like platelets, plasma and red blood cells can be avoided.

Participants will be given one of the two FDA-approved blood products.

DETAILED DESCRIPTION:
Immediately replacing fibrinogen in perioperative bleeding patients with acquired fibrinogen deficiency improves outcomes. The product that is primarily used for fibrinogen replacement in the US, cryoprecipitate (cryo), must be stored frozen and expires six hours after thawing, resulting in a delay in transfusion of approximately 50 minutes from the time it is ordered, as well as unnecessary transfusion of more readily available but not indicated blood components that are transfused while the patients waits for cryo . A modified version of the product, pathogen reduced (PR) cryo, is now FDA approved and can be thawed and stored for 5 days, allowing the product to be available immediately when needed. In this quality improvement study, the investigators will compare the effect that readily available, pre-thawed PR cryo has on transfusion practice in cardiovascular and liver transplant patients who receive PR cryo versus those who receive traditional cryo by randomizing cryo transfusions in the blood bank by month to all cryo or all PR cryo. All clinical decisions, including the need for cryo, and laboratory testing will occur per standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients undergoing cardiovascular surgery or liver transplant who receive cryo during surgery during the two year study period.
2. Cardiovascular surgery includes the following procedures:

   1. coronary artery bypass grafting
   2. valve repair or replacement
   3. open thoracic aortic and thoracoabdominal aortic surgery
   4. atrial or ventricular septal defects
   5. ventricular assist device implantation or revision
   6. or any combination of the above.

Exclusion Criteria:

1. Patients who do not receive any cryo product in the OR
2. Patients who are not cardiovascular surgery or liver transplant patients
3. Cardiac transplantation surgery
4. Patients who receive a product in error within either the cryo time period or the PR cryo time period. For example, PR cryo during a cryo month or cryo during a PR cryo time month.
5. Patients who receive less than 1 pool (5 units) of cryo
6. Pediatric patients (less than 18 years of age).
7. Patients who received both PR cryo and traditional cryo
8. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2025-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Cushing, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York-Presbyterian Hospital/Weill Cornell Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arnup SJ, Forbes AB, Kahan BC, Morgan KE, McKenzie JE. Appropriate statistical methods were infrequently used in cluster-randomized crossover trials. J Clin Epidemiol. 2016 Jun;74:40-50. doi: 10.1016/j.jclinepi.2015.11.013. Epub 2015 Nov 26. PMID 26633599
- [Background] Saland LC. Effects of reserpine administration on the fine structure of the rat pars intermedia. Cell Tissue Res. 1978 Nov 9;194(1):115-23. doi: 10.1007/BF00209237. PMID 719724
- [Background] Cushing MM, Fitzgerald MM, Harris RM, Asmis LM, Haas T. Influence of cryoprecipitate, Factor XIII, and fibrinogen concentrate on hyperfibrinolysis. Transfusion. 2017 Oct;57(10):2502-2510. doi: 10.1111/trf.14259. Epub 2017 Jul 21. PMID 28734018
- [Background] Cushing MM, Haas T, Karkouti K, Callum J. Which is the preferred blood product for fibrinogen replacement in the bleeding patient with acquired hypofibrinogenemia-cryoprecipitate or fibrinogen concentrate? Transfusion. 2020 Jun;60 Suppl 3:S17-S23. doi: 10.1111/trf.15614. Epub 2020 Jun 1. PMID 32478877
- [Background] Fenderson JL, Meledeo MA, Rendo MJ, Peltier GC, McIntosh CS, Davis KW, Corley JB, Cap AP. Hemostatic characteristics of thawed, pooled cryoprecipitate stored for 35 days at refrigerated and room temperatures. Transfusion. 2019 Apr;59(S2):1560-1567. doi: 10.1111/trf.15180. PMID 30980741
- [Background] Bulkley GB, Wheaton LG, Strandberg JD, Zuidema GD. Assessment of small intestinal recovery from ischemic injury after segmental, arterial, venous, and arteriovenous occlusion. Surg Forum. 1979;30:210-3. No abstract available. PMID 538597
- [Background] Hsien S, Dayton JD, Chen D, Stock A, Bacha E, Cushing MM, Nellis ME. Hemostatic efficacy of pathogen-reduced platelets in children undergoing cardiopulmonary bypass. Transfusion. 2022 Feb;62(2):298-305. doi: 10.1111/trf.16768. Epub 2021 Dec 13. PMID 34904250
- [Background] Lokhandwala PM, O'Neal A, Patel EU, Brunker PAR, Gehrie EA, Zheng G, Kickler TS, Ness PM, Tobian AAR. Hemostatic profile and safety of pooled cryoprecipitate up to 120 hours after thawing. Transfusion. 2018 May;58(5):1126-1131. doi: 10.1111/trf.14550. Epub 2018 Feb 25. PMID 29479708
- [Background] Thomson C, Sobieraj-Teague M, Scott D, Duncan E, Abraham S, Roxby D. Extending the post-thaw viability of cryoprecipitate. Transfusion. 2021 May;61(5):1578-1585. doi: 10.1111/trf.16366. Epub 2021 Mar 17. PMID 33728705
- [Derived] Cushing MM, Cohen T, Fitzgerald MM, Rand S, Sinfort A, Chen D, Keltner N, Ong S, Parra P, Benabdessadek D, Jimenez A, Haas T, Lau C, Girardi NI, DeSimone RA. Trial Of Pathogen-reduced Cryoprecipitate vs. Cryoprecipitated AHF to Lower Operative Transfusions (TOP-CLOT): study protocol for a single center, prospective, cluster randomized trial. Trials. 2024 Sep 27;25(1):625. doi: 10.1186/s13063-024-08398-x. PMID 39334317

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: cryo transfusions
Groups:
- Patients Given Traditional Cryo: These are all liver transplant and cardiothoracic (LT and CT) patients that will be given Traditional Cryo based on the randomization protocol. The blood bank will be randomized by to use either PR Cryo or Traditional Cryo for the entire month for all patients with a Cryo order. The patients included in this arm received Traditional Cryo during a month in which the blood bank was randomized to use Traditional Cryo. The months in which the blood bank was assigned to use Traditional Cryo are as follows: Period 1: Month 1, Period 4: Month 4, Period 5: Month 5, Period 7: Month 7, Period 10: Month 10, and Period 12: Month 12.
- Patients Given PR Cryo: These are all liver transplant and cardiothoracic (LT and CT) patients that will be given PR Cryo based on the randomization protocol. The blood bank will be randomized by to use either PR Cryo or Traditional Cryo for the entire month for all patients with a Cryo order. The patients included in this arm received PR Cryo during a month in which the blood bank was randomized to use PR Cryo. The months in which the blood bank was assigned to use PR Cryo are as follows: Period 2: Month 2, Period 3: Month 3, Period 6: Month 6, Period 8: Month 8, Period 9: Month 9, Period 11: Month 11.
Period: Month 1 (Traditional Cryo)
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Started | 20; 50 cryo transfusions | 0; 0 cryo transfusions
Completed | 20; 50 cryo transfusions | 0; 0 cryo transfusions
Not Completed | 0; 0 cryo transfusions | 0; 0 cryo transfusions
Period: Month 2 (PR Cryo)
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Started | 0; 0 cryo transfusions | 20; 45 cryo transfusions
Completed | 0; 0 cryo transfusions | 20; 45 cryo transfusions
Not Completed | 0; 0 cryo transfusions | 0; 0 cryo transfusions
Period: Month 3 (PR Cryo)
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Started | 0; 0 cryo transfusions | 17; 43 cryo transfusions
Completed | 0; 0 cryo transfusions | 17; 43 cryo transfusions
Not Completed | 0; 0 cryo transfusions | 0; 0 cryo transfusions
Period: Month 4 (Traditional Cryo)
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Started | 20; 42 cryo transfusions | 0; 0 cryo transfusions
Completed | 20; 42 cryo transfusions | 0; 0 cryo transfusions
Not Completed | 0; 0 cryo transfusions | 0; 0 cryo transfusions
Period: Month 5 (Traditional Cryo)
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Started | 20; 51 cryo transfusions | 0; 0 cryo transfusions
Completed | 20; 51 cryo transfusions | 0; 0 cryo transfusions
Not Completed | 0; 0 cryo transfusions | 0; 0 cryo transfusions
Period: Month 6 (PR Cryo)
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Started | 0; 0 cryo transfusions | 19; 40 cryo transfusions
Completed | 0; 0 cryo transfusions | 19; 40 cryo transfusions
Not Completed | 0; 0 cryo transfusions | 0; 0 cryo transfusions
Period: Month 7 (Traditional Cryo)
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Started | 23; 41 cryo transfusions | 0; 0 cryo transfusions
Completed | 23; 41 cryo transfusions | 0; 0 cryo transfusions
Not Completed | 0; 0 cryo transfusions | 0; 0 cryo transfusions
Period: Month 8 (PR Cryo)
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Started | 0; 0 cryo transfusions | 15; 28 cryo transfusions
Completed | 0; 0 cryo transfusions | 15; 28 cryo transfusions
Not Completed | 0; 0 cryo transfusions | 0; 0 cryo transfusions
Period: Month 9 (PR Cryo)
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Started | 0; 0 cryo transfusions | 19; 44 cryo transfusions
Completed | 0; 0 cryo transfusions | 19; 44 cryo transfusions
Not Completed | 0; 0 cryo transfusions | 0; 0 cryo transfusions
Period: Month 10 (Traditional Cryo)
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Started | 10; 21 cryo transfusions | 0; 0 cryo transfusions
Completed | 10; 21 cryo transfusions | 0; 0 cryo transfusions
Not Completed | 0; 0 cryo transfusions | 0; 0 cryo transfusions
Period: Month 11 (PR Cryo)
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Started | 0; 0 cryo transfusions | 13; 38 cryo transfusions
Completed | 0; 0 cryo transfusions | 13; 38 cryo transfusions
Not Completed | 0; 0 cryo transfusions | 0; 0 cryo transfusions
Period: Month 12 (Traditional Cryo)
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Started | 12; 35 cryo transfusions | 0; 0 cryo transfusions
Completed | 12; 35 cryo transfusions | 0; 0 cryo transfusions
Not Completed | 0; 0 cryo transfusions | 0; 0 cryo transfusions

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo | Total
Number analyzed (Participants) | 105 | 103 | 208
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (14) | 61 (14) | 61 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 41 | 80
  Male | 66 | 62 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 1 | 15
  Unknown or Not Reported | 91 | 102 | 193
Region of Enrollment [Number; unit: participants]
  United States | 105 | 103 | 208
ASA Score [Mean (Standard Deviation); unit: Score on a scale] — The ASA Score (American Society of Anesthesiologists Physical Status Classification System) assesses a patient's preoperative health. Scores range from 1 to 6. Score 1 indicates healthy; Score 2 indicates mild systemic disease; Score 3 indicates severe systemic disease; Score 4 indicates disease that is a constant threat to life; Score 5 indicates a moribund patient not expected to survive without surgery; Score 6 indicates a brain-dead patient whose organs are being removed for donor purposes.
  Score on a scale | 3.8 (0.51) | 3.8 (0.43) | 3.8 (0.47)

OUTCOME MEASURES:

1. Primary Outcome: Total Number of RBCs Used Over Admission
Description: RBCs used over admission
Time Frame: Within the first 30 days after surgery.
Measure: Mean (Standard Deviation); unit: RBC Units
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 105 | 103
RBC Units | 5.8 (6.5) | 6.7 (7.2)

2. Primary Outcome: Total Number of Platelets Used Over Admission
Description: Plts used over admission
Time Frame: Within the first 30 days after surgery.
Measure: Mean (Standard Deviation); unit: platelet units
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 105 | 103
platelet units | 2.1 (3.1) | 2.1 (2.0)

3. Primary Outcome: Total Number of Plasma Used Over Admission
Description: All units over admission
Time Frame: Within the first 30 days after surgery.
Measure: Mean (Standard Deviation); unit: plasma units
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 105 | 103
plasma units | 2.7 (4.6) | 3.4 (6.0)

4. Secondary Outcome: Number of Cryo Units Used Perioperatively
Description: All products within 3 days
Time Frame: 3 days post procedure
Measure: Mean (Standard Deviation); unit: cryo units
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 105 | 103
cryo units | 2.3 (1.7) | 2.3 (1.6)

5. Secondary Outcome: Number of RBCs Used Perioperatively
Description: Number of RBC units transfused during perioperative period
Time Frame: 3 days post procedure
Measure: Mean (Standard Deviation); unit: RBC units
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 105 | 103
RBC units | 4.6 (5.6) | 5.9 (6.6)

6. Secondary Outcome: Number of Plasma Used Perioperatively
Time Frame: 3 days post procedure
Measure: Mean (Standard Deviation); unit: plasma units
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 105 | 103
plasma units | 2.6 (4.6) | 3.4 (6.01)

7. Secondary Outcome: Number of Platelets Used Perioperatively
Description: Number of platelet units transfused during perioperative period
Time Frame: 3 days post procedure
Measure: Mean (Standard Deviation); unit: platelet units
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 105 | 103
platelet units | 1.8 (1.7) | 2.0 (1.8)

8. Secondary Outcome: Time From Operating Room (OR) Start Time to Start of Cryo Transfusion
Time Frame: procedure (Time from OR start time to start of cryo transfusion)
Population: Only the cardiac population was included for this analysis. The data was not available for liver transplant patients, so liver transplant patients were excluded from the analysis.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 86 | 84
minutes | 366 [309 to 425] | 367 [324 to 416]

9. Secondary Outcome: Time From Cryo Order to Start of Transfusion
Description: Time to cryo order time to start of cryo transfusion
Time Frame: procedure (Time from cryo order to start of transfusion)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 105 | 103
minutes | 128.3 (200.7) | 88.5 (99.8)

10. Secondary Outcome: Number of Cryo Units Wasted by Blood Bank
Description: This captures the Cryoprecipitate units discarded.
Time Frame: Daily, up to approximately 24 months
Population: The blood bank, which is required to follow its standard operating procedures, was not able to document wastage in a way which allowed the investigators to accurately attribute wastage to a specific arm of the study. Therefore, wastage could not be accurately calculated as intended in the study protocol.
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Pre Transfusion FIBTEM Amplitude 10 Min After Start of Clot Formation
Description: FIBTEM before transfusion, if anesthesiologist orders it. FIBTEM is a point of care laboratory test measuring fibrinogen contribution to a clot. It is part of ROTEM testing and helps providers determine if patients need fibrinogen supplementation during surgical bleeding.
Time Frame: Variable, but it is generally available within 15 minutes of the start of ROTEM testing.
Population: Data for all participants was not available because pre-transfusion FIBTEMs were not clinically ordered for all participants by the treating anesthesiologists. Only participants with pre-transfusion FIBTEMs available were included in this analysis.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 95 | 94
mm | 9.6 (6.8) | 8.3 (4.2)

12. Secondary Outcome: Post Transfusion FIBTEM Amplitude at 10 Min After Start of Clot Formation
Description: FIBTEM after transfusion, if anesthesiologist orders it. FIBTEM is a point of care laboratory test measuring fibrinogen contribution to a clot. It is part of ROTEM testing and helps providers determine if patients need fibrinogen supplementation during surgical bleeding.
Time Frame: Variable, but it is generally available within 15 minutes of the start of ROTEM testing.
Population: Data were not available nor collected for this measure because anesthesiologists do not routinely order this for the investigators to have been able to collect it.
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Maximum Clot Firmness (MCF)
Description: The maximum strength of a clot as determined by ROTEM testing.
Time Frame: Variable, but it is generally available within 1 hour of the start of ROTEM testing.
Population: Data for MCF were not collected since clinical decisions are not made based on this value as the measure assumed. As such, there are no data to report. Clinical decisions were made based on A10 (the clot amplitude measured 10 minutes after clot formation start), not the maximum clot firmness (MCF). As A10 was not a pre-specified measure for this protocol, there are no data to report. Data will never be collected for this Outcome Measure.
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Pre-transfusion Fibrinogen Level
Description: The fibrinogen measurement before cryoprecipitate is transfused.
Time Frame: During surgery, within 3 hours of specimen receipt by laboratory.
Population: Some data were not collected for this measure because anesthesiologists did not routinely order this test.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 10 | 9
mg/dL | 145 (68) | 191 (33)

15. Secondary Outcome: Highest Fibrinogen Level Within 24 Hours
Time Frame: Within 24 hours after surgery
Population: Some data were not collected for this measure because anesthesiologists did not always order this test.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 100 | 100
mg/dL | 210 (53) | 212 (46)

16. Secondary Outcome: Lowest Fibrinogen Level Within 24 Hours
Time Frame: Within 24 hours after surgery
Population: Some data were not collected for this measure because anesthesiologists did not always order this test.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 100 | 100
mg/dL | 194.5 (51.0) | 199.89 (44.3)

17. Secondary Outcome: Cumulative Volume in Drains After Surgery (e.g., Chest Tube for CV Surgery) at the Time of Removal
Description: The cumulative volume in drains after surgery (e.g., chest tube for CV surgery) at the time of drain removal
Time Frame: Up to approximately 3 days
Population: This data were not available for collection in the electronic health record as intended by the investigators, as the data were not clinically documented. Therefore, the cumulative volume in drains after surgery could not be reported as intended in the study protocol.
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Volume in Drains (Chest Tube for CV Surgery)
Time Frame: At 24 hours after surgery
Population: Only the cardiac population was included for this analysis. The clinical parameter is not applicable to liver transplant patients, so liver transplant patients were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: mLs
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 85 | 83
mLs | 897 (810) | 749 (496)

19. Secondary Outcome: Time From End of Bypass Pump for CV Surgery
Time Frame: Until end of surgery
Population: Only for cardiac surgery patients. Liver transplant patients are not on bypass.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 86 | 84
hours | 2.75 [2.32 to 3.27] | 2.73 [2.46 to 3.22]

20. Secondary Outcome: Length of Stay in OR
Description: Operating room length of stay
Time Frame: Duration of time in operating room
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 105 | 103
minutes | 522 (124) | 534 (118)

21. Secondary Outcome: Length of Stay in ICU
Description: Participant length of stay in ICU setting
Time Frame: During hospitalization, approximately 5 days to 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 105 | 103
days | 8.1 (11.8) | 6.9 (8.6)

22. Secondary Outcome: Length of Stay in Hospital
Description: Overall length of stay in hospital
Time Frame: During hospitalization, approximately 5 days to 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 105 | 103
days | 12.0 (9.4) | 10.9 (10.1)

23. Secondary Outcome: Need for Ventilator
Time Frame: During hospitalization, approximately 5 days to 30 days
Population: Not all values available in the electronic health record.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 100 | 98
Participants | 99 | 96

24. Secondary Outcome: Time on Ventilator
Description: If participant was on ventilator, amount of time spent on ventilator
Time Frame: During hospitalization, approximately 5 days to 30 days
Population: Not all values available in the electronic health record.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 99 | 96
days | 2.4 (4.9) | 2.6 (6.3)

25. Secondary Outcome: Overall Cost of Cryo vs PR Cryo, When Factoring Wastage
Description: Cost of traditional cryoprecipitate compared to PR Cryoprecipitate.
Time Frame: Daily, approximately 24 months
Population: Not available due to unavailable confidential contractual information that would be needed to calculate cost. The contract between the blood suppliers and hospital is confidential, and therefore the investigators were not able to report on cost-related factors as intended in the study protocol. Data will never be collected for this Outcome Measure.
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Number of Participants That Experienced an Adverse Event of Fever
Description: All participants that experience fevers that occur during the time frame
Time Frame: Within 5 days of surgery start time
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 105 | 103
Participants | 16 | 14

27. Secondary Outcome: Number of Participants That Experienced an Adverse Event of Infection
Description: All participants that experience infections that occur during the time frame
Time Frame: Within 5 days of surgery start time
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 105 | 103
Participants | 6 | 4

28. Secondary Outcome: Number of Participants That Experienced an Adverse Event of Transfusion Reaction.
Description: All participants that experience transfusion reactions that occur during the time frame
Time Frame: Within 5 days of surgery start time
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 105 | 103
Participants | 0 | 0

29. Secondary Outcome: Fibrinogen Level
Description: Fibrinogen level most proximal to the end of surgery
Time Frame: Most proximal to end of procedure
Population: Fibrinogen was not ordered by provider for every participant
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
Number analyzed (Participants) | 101 | 101
mg/dL | 197 (52) | 201 (38)

ADVERSE EVENTS:
Time Frame: Serious adverse events: 5 days post-procedure. All cause-mortality: 30 days or discharge from hospital, whichever occurred first.
Description: Serious adverse events collected included transfusion reactions. Adverse events collected included fevers and infections. Data were collected using automated scripts with Structured Query Language (SQL) queries of the hospital's centralized data warehouse. Adverse events were assessed weekly by the study team via video conference.
Arm/Group | Patients Given Traditional Cryo | Patients Given PR Cryo
All-Cause Mortality (participants affected / at risk) | 5/105 | 2/103
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/103
Other Adverse Events (participants affected / at risk) | 18/105 | 17/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Given Traditional Cryo (N=105) | Patients Given PR Cryo (N=103)
Transfusion Reactions (Blood and lymphatic system disorders) | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Given Traditional Cryo (N=105) | Patients Given PR Cryo (N=103)
Infection (Infections and infestations) | 6 (6) | 4 (4)
Fever (Infections and infestations) | 16 (16) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/24/NCT05711524/Prot_SAP_000.pdf